CLINICAL TRIAL: NCT00000112
Title: Prevalence of Carbohydrate Intolerance in Lean and Obese Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR06022-0029; M01RR006022 (NIH)
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Obesity; Glucose Intolerance; Diabetes; Acanthosis Nigricans
MeSH Terms: conditions — Obesity; Glucose Intolerance; Diabetes Mellitus; Acanthosis Nigricans

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The prevalence of obesity in children is reaching epidemic proportions. Excess adiposity is more than just a cosmetic problem, having substantial metabolic consequences. Insulin resistance, hyperinsulinemia, impaired glucose tolerance, and frank diabetes are often seen in obese children. In this study the prevalence of impaired glucose (carbohydrate) tolerance in lean children with a family history of diabetes and obese children with acanthosis nigricans with or without a family history of diabetes mellitus will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Obesity: BM +/- 95% for age general good health

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University School of Medicine, Pediatric Endocrinology, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Halloun R, Galderisi A, Caprio S, Weiss R. Adipose Tissue Insulin Resistance Is Not Associated With Changes in the Degree of Obesity in Children and Adolescents. J Clin Endocrinol Metab. 2023 Apr 13;108(5):1053-1060. doi: 10.1210/clinem/dgac700. PMID 36469736
- [Derived] Halloun R, Galderisi A, Caprio S, Weiss R. Lack of Evidence for a Causal Role of Hyperinsulinemia in the Progression of Obesity in Children and Adolescents: A Longitudinal Study. Diabetes Care. 2022 Jun 2;45(6):1400-1407. doi: 10.2337/dc21-2210. PMID 35235641
- [Derived] Ricke J, Klumpen HJ, Amthauer H, Bargellini I, Bartenstein P, de Toni EN, Gasbarrini A, Pech M, Peck-Radosavljevic M, Popovic P, Rosmorduc O, Schott E, Seidensticker M, Verslype C, Sangro B, Malfertheiner P. Impact of combined selective internal radiation therapy and sorafenib on survival in advanced hepatocellular carcinoma. J Hepatol. 2019 Dec;71(6):1164-1174. doi: 10.1016/j.jhep.2019.08.006. Epub 2019 Aug 14. PMID 31421157